CLINICAL TRIAL: NCT02314195
Title: A Randomized Clinical Trial of Music Therapy as an Adjunct to Standard Treatment for Obsessive Compulsive Disorder and Co-morbid Anxiety and Depression in Iran
Brief Title: Music Therapy in Obsessive Compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamic Azad University, Marvdasht (Other)
Responsible Party: Principal Investigator, Shahrzad Shirani, Shahrzad Shirani Bidabadi, M.S.c, Islamic Azad University, Marvdasht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2172719
Record Dates: First submitted 2014-11-27; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Obsessive-Compulsive Disorder; Anxiety; Depression
Keywords: Obsessive Compulsive Disorder; Music Therapy/methods; Combined Modality Therapy; Anxiety Disorders/therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Anxiety Disorders; Depression | interventions — Selective Serotonin Reuptake Inhibitors; Drug Therapy; Cognitive Behavioral Therapy; Psychotherapy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard treatment + music therapy (Active Comparator): Selective serotonin re-uptake inhibitor plus cognitive behavioral therapy. Music therapy encompassing 12 half-hour sessions of therapist-supervised receptive music therapy scheduled over four weeks
  Interventions: Drug: Selective serotonin re-uptake inhibitor; Behavioral: Cognitive Behavioral Therapy; Other: Music therapy
- Standard treatment only (Active Comparator): Selective serotonin re-uptake inhibitor plus cognitive behavioral therapy.
  Interventions: Drug: Selective serotonin re-uptake inhibitor; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Selective serotonin re-uptake inhibitor — A medication of selective serotonin re-uptake inhibitor (SSRI) family, Behavioral. The type and dosage of the medication was decided by the treating psychiatrist.
  Other Names: Pharmacotherapy
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy for obsessive compulsive disorder carried out by a psychologist.
  Other Names: Psychotherapy
Other: Music therapy — 12 sessions of 30-minute individual-based receptive music therapy, supervised by the treating psychiatrist.
  Other Names: Receptive music therapy
  Arms: Standard treatment + music therapy

SUMMARY:
Previous studies have highlighted the potential therapeutic benefits of receptive individual music therapy as an adjunct to standard care, in a variety of psychiatric ailments including mood and anxiety disorders. However, the role of music in the treatment of obsessive compulsive disorder have not been investigated to date. The present study therefore aimed to investigate the efficacy of music therapy as an adjunct to standard treatment, on obsessions in patients with treatment-naïve OCD. Moreover, given the fact that a significant proportion of patients with OCD have other comorbid mood or anxiety disorders, the question of whether therapeutic benefits of music could be expanded to also affect concurrent depressive and anxiety symptoms was explored.

ELIGIBILITY:
Inclusion Criteria:

* were at least 18 years or older;
* had axis I diagnosis of OCD according to the criteria delineated by the diagnostic and statistical manual of mental disorders - fourth edition diagnosed by an experienced psychiatrist
* had not received treatment previously for the disorder
* agreed to partake in the study

Exclusion Criteria:

* refused to partake in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Obsession (Maudsley Obsessive-Compulsive Inventory) | 1 month
  Post-intervention scores on Maudsley Obsessive-Compulsive Inventory

SECONDARY OUTCOMES:
Obsession subtype (Maudsley Obsessive-Compulsive Inventory sub-types) | 1 month
  Post-intervention scores on Maudsley Obsessive-Compulsive Inventory sub-types
Anxiety symptoms (Beck Anxiety Inventory) | 1 month
  Post-intervention scores on Beck Anxiety Inventory
Depressive symptoms (Beck Depression Inventory - Short Form) | 1 month
  Post-intervention scores on Beck Depression Inventory - Short Form

CONTACTS AND LOCATIONS:
Locations (1):
- Shariati Hospital, Isfahan, Isfahan, Iran